CLINICAL TRIAL: NCT02782884
Title: A Prospective Study of Post-operative Opioid Use in General Surgical Patients
Brief Title: A Prospective Study of Post-operative Opioid Use in General Surgery Patients
Acronym: GSopioids
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Richard J. Barth,Jr., Staff Physician, General Surgery, Dartmouth-Hitchcock Medical Center
Other Study IDs: D16112
Record Dates: First submitted 2016-05-22; First posted 2016-05-25 (Estimated); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: Pain
Keywords: post-operative pain
MeSH Terms: conditions — Pain; Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Outpatient general surgery operation: Patients undergoing outpatient general surgical operations They will be given a specified number of narcotic pills based on our retrospective analysis of patient post-operative opioid use
- Inpatient general surgical patients: Inpatients who are being discharged They will be given a specified number of narcotic pills based on the number of pills they took in the 24 hrs prior to discharge

SUMMARY:
Patients undergoing approximately 10 common outpatient general surgical operations will be given a narcotic prescription for a specified number of pills.

Inpatients who are about to be discharged after surgery or trauma will be given narcotic prescriptions for a specified number of pills. Patients will be given a patient report form which they will use to record the number of pills they take each day and their daily pain score on a scale of 0-10.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* undergoing one of 9 elective outpatient operations: partial mastectomy, partial mastectomy and sentinel node biopsy, melanoma wide excision and sentinel node excision, thyroidectomy, parathyroidectomy, open inguinal hernia repair, laparoscopic inguinal hernia repair, laparoscopic cholecystectomy OR
* an inpatient on the general surgery service who took at least one oral narcotic

Exclusion Criteria:

* allergic to all narcotics
* chronic opioid use
* history of opioid or benzodiazepine abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: >= 18 years of age undergoing one of 9 elective outpatient operations: partial mastectomy, partial mastectomy and sentinel node biopsy, melanoma wide excision and sentinel node excision, thyroidectomy, parathyroidectomy, open inguinal hernia repair, laparoscopic inguinal hernia repair, laparoscopic cholecystectomy OR an inpatient on the general surgery service who took at least one oral narcotic in the 24 hrs prior to discharge
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2017-08-04 (Actual); Study Completion 2017-08-16 (Actual)

PRIMARY OUTCOMES:
number of pills to satisfy 80% of patients opioid needs | 1 yr

SECONDARY OUTCOMES:
proportion of patients requiring narcotic refills when specified number of pills is given | 1 year
patient pain level, daily | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Barth, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center

IPD SHARING:
Plan to Share IPD: No